CLINICAL TRIAL: NCT02487160
Title: Clinical Evaluation of the Lenstec SBL-3 Multifocal Intraocular Lens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lenstec Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBL-INI-02-13
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Cataracts; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Intervention Model Description: SBL-3 multifocal intraocular lens
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBL-3 multifocal intraocular lens (Experimental): The SBL-3 intraocular lens will be implanted after the cataractous natural lens has been removed, in those patients randomized into this group
  Interventions: Device: SBL-3 multifocal intraocular lens
- Control monofocal intraocular lens (Active Comparator): The Control intraocular lens will be implanted after the cataractous natural lens has been removed, in those patients randomized into this group
  Interventions: Device: Control monofocal intraocular lens

INTERVENTIONS:
Device: SBL-3 multifocal intraocular lens — The SBL-3 intraocular lens will be implanted after the cataractous natural lens has been removed, in those patients randomized into this group
  Arms: SBL-3 multifocal intraocular lens
Device: Control monofocal intraocular lens — The Control intraocular lens will be implanted after the cataractous natural lens has been removed, in those patients randomized into this group
  Arms: Control monofocal intraocular lens

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the SBL-3 intraocular lens.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety (adverse events) and performance (visual acuity, spectacle independence) of the SBL-3 intraocular lens.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 22 years of age, of any race and either gender
2. Operable, age related cataract grade in both eyes
3. Patients who require an intraocular lens (IOL) power in the range of 15 D - 30 D only
4. Able to comprehend and sign a statement of informed consent
5. Calculated lens power within the available supply range
6. Planned cataract removal by phacoemulsification
7. Potential postoperative visual acuity of 0.2 Logarithm of the Minimum Angle of Resolution (logMAR) or better in both eyes
8. In good general and ocular health
9. Patients with preoperative astigmatism ≤1.0 D Note: Corneal incisions made to reduce astigmatism will not be allowed during the course of the study.
10. Clear intraocular media other than cataract in study eyes
11. Preoperative Best Corrected Distance Visual Acuity (BCDVA) worse than 0.2 logMAR
12. The subject must be able to undergo second eye surgery between 7 days and 30 days of the first eye surgery
13. Able to competently complete testing
14. Willing and able to attend study visits

Exclusion Criteria:

1. Previous intraocular surgery
2. Preoperative photopic pupil size of < 2.75 mm
3. Previous corneal refractive surgery
4. Any inflammation or edema (swelling) of the cornea
5. Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders ) that are predicted to cause future acuity losses to a level worse than 0.2 logMAR
6. Subjects who may reasonably be expected to require a secondary surgical intervention at any time during the study (other than neodymium-doped yttrium aluminium garnet (nd:YAG) capsulotomy)
7. Amblyopia
8. Clinically significant ptosis
9. Clinically severe corneal dystrophy (eg., epithelial, stromal, or endothelial dystrophy), keratitis, keratoconjunctivitis, keratouveitis, keratopathy, or kerectasia
10. Diabetic Retinopathy
11. Extremely shallow anterior chamber, not due to swollen cataract
12. Microphthalmia
13. Previous retinal detachment
14. Previous corneal transplant
15. Severe dry eye
16. Recurrent severe anterior or posterior segment inflammation of unknown etiology
17. Systemic medications that may confound the outcome or increase the risk to the subject in the opinion of the Investigator [tamsulosin hydrochloride (Flomax) or other medications with similar side effects (floppy iris syndrome)]
18. Rubella or traumatic cataract
19. Iris neovascularization
20. Glaucoma (medically controlled or uncontrolled)
21. Aniridia
22. Chronic severe uveitis
23. Optic nerve atrophy
24. Corneal decompensation
25. Greater than 1.0 D of astigmatism
26. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.)
27. Pseudoexfoliation syndrome
28. Iris atrophy
29. Pupil abnormalities (e.g., corectopia)
30. Aniseikonia
31. An acute or chronic disease or illness that may confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness)
32. Pregnant, lactating, or planning to become pregnant during the course of the trial Note: Subjects who become pregnant during the study will not be discontinued; however, data may be excluded from the effectiveness analyses because pregnancy can alter refraction and visual acuity results.
33. Participation in another clinical trial within 30 days of study start

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2015-08; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
photopic, distance corrected, monocular near visual acuity | 1 year following implantation
  a measure of near vision
presence or absence of adverse events | 1 year following implantation
  presence or absence of adverse events
photopic, distance corrected, monocular intermediate visual acuity | 1 year following implantation
  a measure of intermediate vision
photopic, best corrected, monocular distance visual acuity | 1 year following implantation
  a measure of distance vision

SECONDARY OUTCOMES:
Proportion of subjects who are independent of spectacles | 1 year following implantation
  a measure of the independence from spectacles

CONTACTS AND LOCATIONS:
Overall Officials: Blake Harris, Study Director — Lenstec Inc
Locations (13):
- United States (13):
  - Eye Center South, Dothan, Alabama
  - Shepard Eye Center, Santa Maria, California
  - Cape Coral Eye Center, Cape Coral, Florida
  - Eye Centers of Florida, Fort Myers, Florida
  - Newsom Eye & Laser Center, Sebring, Florida
  - Family Eye Centers, Willmar, Minnesota
  - The Eye Center of Central PA, Allenwood, Pennsylvania
  - Eye Care Specialists, Kingston, Pennsylvania
  - Carolina Eyecare Physicians, Mt. Pleasant, South Carolina
  - Loden Vision Center, Goodlettsville, Tennessee
  - Kleiman/Evangelista Eye Center, Arlington, Texas
  - Whitsett Vision Group, Houston, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shields AL, Galipeau N, Litcher-Kelly L, Moreno-Koehler A, Chacko J. The patient reported intraocular lens questionnaire (PR-ILQ): content validity, psychometric performance, and use in a regulated clinical trial to evaluate safety and effectiveness outcomes. J Patient Rep Outcomes. 2025 Dec 12;9(1):142. doi: 10.1186/s41687-025-00968-0. PMID 41385130